CLINICAL TRIAL: NCT05106153
Title: A Single-Dose, Double-Blind, Placebo-Controlled, Randomized, Crossover Study to Determine the Abuse Potential of Single Oral Dose of Seltorexant Compared To Suvorexant and Zolpidem
Brief Title: A Study to Determine the Abuse Potential of Seltorexant Compared to Suvorexant and Zolpidem
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR109099; 42847922MDD1017 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-10-21; First posted 2021-11-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy Non-dependent, Recreational Sedative Users; Abuse Potential
MeSH Terms: interventions — suvorexant; Zolpidem; seltorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Qualification Phase: Treatment Sequence YXZ (Experimental): Participants will receive a single oral dose of suvorexant (Treatment Y) in qualification period 1, followed by single oral dose of placebo (Treatment X) in qualification period 2 and then single oral dose of zolpidem (Treatment Z) in qualification period 3 on Day 1 during each qualification phase. Each treatment will be separated by washout of at least 3 days.
  Interventions: Drug: Suvorexant; Drug: Zolpidem; Drug: Placebo
- Qualification Phase: Treatment Sequence ZYX (Experimental): Participants will receive Treatment Z in qualification period 1, followed by Treatment Y in qualification period 2, and then Treatment X in qualification period 3 on Day 1 during each qualification phase. Each treatment will be separated by washout of at least 3 days.
  Interventions: Drug: Suvorexant; Drug: Zolpidem; Drug: Placebo
- Qualification Phase: Treatment Sequence XZY (Experimental): Participants will receive Treatment X in qualification period 1, followed by Treatment Z in qualification period 2, and then Treatment Y in qualification period 3 on Day 1 during each qualification phase. Each treatment will be separated by washout of at least 3 days.
  Interventions: Drug: Suvorexant; Drug: Zolpidem; Drug: Placebo
- Qualification Phase: Treatment Sequence YZX (Experimental): Participants will receive Treatment Y in qualification period 1, followed by Treatment Z in qualification period 2, and then Treatment X in qualification period 3 on Day 1 during each qualification phase. Each treatment will be separated by washout of at least 3 days.
  Interventions: Drug: Suvorexant; Drug: Zolpidem; Drug: Placebo
- Qualification Phase: Treatment Sequence ZXY (Experimental): Participants will receive Treatment Z in qualification period 1, followed by Treatment X in qualification period 2, and then Treatment Y in qualification period 3 on Day 1 during qualification phase. Each treatment will be separated by washout of at least 3 days.
  Interventions: Drug: Suvorexant; Drug: Zolpidem; Drug: Placebo
- Qualification Phase: Treatment Sequence XYZ (Experimental): Participants will receive Treatment X in qualification period 1, followed by Treatment Y in qualification period 2, and then Treatment Z in qualification period 3 on Day 1 during each qualification phase. Each treatment will be separated by washout of at least 3 days.
  Interventions: Drug: Suvorexant; Drug: Zolpidem; Drug: Placebo
- Treatment Phase: Treatment Sequence ABFCED (Experimental): Participants will receive a single oral dose of placebo (Treatment A) in treatment period 1, followed by single oral dose of suvorexant (Treatment B) in treatment period 2, single oral Dose 3 of seltorexant (Treatment F) in treatment period 3, single oral dose of zolpidem (Treatment C) in treatment period 4, single oral Dose 2 of seltorexant (Treatment E) in treatment period 5 and then a single oral Dose 1 of seltorexant (Treatment D) in treatment period 6 on Day 1 during each treatment phase. Each treatment will be separated by washout of at least 5 days.
  Interventions: Drug: Suvorexant; Drug: Zolpidem; Drug: Seltorexant; Drug: Placebo
- Treatment Phase: Treatment Sequence BCADFE (Experimental): Participants will receive Treatment B in treatment period 1, followed by Treatment C in treatment period 2, Treatment A in treatment period 3, Treatment D in treatment period 4, Treatment F in treatment period 5 and then Treatment E in treatment period 6 on Day 1 during each treatment phase. Each treatment will be separated by washout of at least 5 days.
  Interventions: Drug: Suvorexant; Drug: Zolpidem; Drug: Seltorexant; Drug: Placebo
- Treatment Phase: Treatment Sequence CDBEAF (Experimental): Participants will receive Treatment C in treatment period 1, followed by Treatment D in treatment period 2, Treatment B in treatment period 3, Treatment E in treatment period 4, Treatment A in treatment period 5 and then Treatment F in treatment period 6 on Day 1 during each treatment phase. Each treatment will be separated by washout of at least 5 days.
  Interventions: Drug: Suvorexant; Drug: Zolpidem; Drug: Seltorexant; Drug: Placebo
- Treatment Phase: Treatment Sequence DECFBA (Experimental): Participants will receive Treatment D in treatment period 1, followed by Treatment E in treatment period 2, Treatment C in treatment period 3, Treatment F in treatment period 4, Treatment B in treatment period 5 and then Treatment A in treatment period 6 on Day 1 during each treatment phase. Each treatment will be separated by washout of at least 5 days.
  Interventions: Drug: Suvorexant; Drug: Zolpidem; Drug: Seltorexant; Drug: Placebo
- Treatment Phase: Treatment Sequence: EFDACB (Experimental): Participants will receive Treatment E in treatment period 1, followed by Treatment F in treatment period 2, Treatment D in treatment period 3, Treatment A in treatment period 4, Treatment C in treatment period 5 and then Treatment B in treatment period 6 on Day 1 during each treatment phase. Each treatment will be separated by washout of at least 5 days.
  Interventions: Drug: Suvorexant; Drug: Zolpidem; Drug: Seltorexant; Drug: Placebo
- Treatment Phase: Treatment Sequence FAEBDC (Experimental): Participants will receive Treatment F in treatment period 1, followed by Treatment A in treatment period 2, Treatment E in treatment period 3, Treatment B in treatment period 4, Treatment D in treatment period 5 and Treatment C in treatment period 6 on Day 1 during each treatment phase. Each treatment will be separated by washout of at least 5 days.
  Interventions: Drug: Suvorexant; Drug: Zolpidem; Drug: Seltorexant; Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant — Suvorexant will be administered orally as per assigned treatment sequence.
Drug: Zolpidem — Zolpidem will be administered orally as per assigned treatment sequence.
Drug: Seltorexant — Seltorexant will be administered orally as per assigned treatment sequence.
  Other Names: JNJ-42847922
  Arms: Treatment Phase: Treatment Sequence ABFCED; Treatment Phase: Treatment Sequence BCADFE; Treatment Phase: Treatment Sequence CDBEAF; Treatment Phase: Treatment Sequence DECFBA; Treatment Phase: Treatment Sequence FAEBDC; Treatment Phase: Treatment Sequence: EFDACB
Drug: Placebo — Placebo will be administered orally as per assigned treatment sequence.

SUMMARY:
The purpose of this study is to evaluate the abuse potential of seltorexant compared to placebo and two active comparators (zolpidem and suvorexant) in non-dependent, recreational sedative users.

ELIGIBILITY:
Inclusion Criteria:

* Be a current, recreational, not physically dependent, drug user
* Participant must be medically stable
* All female participants must have a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening and a negative urine pregnancy test on Day -1 of the qualification phase and on Day -1 of each treatment period of the treatment Phase
* Blood pressure (after the participant is in a sitting position for 5 minutes) between 90 millimeters of mercury (mmHg) and 160 mmHg systolic, inclusive, and no higher than 100 mmHg diastolic at screening and Day -1 prior to qualification phase randomization
* A 12-lead ECG consistent with normal cardiac conduction and function, including: sinus rhythm, pulse rate between 40 and 100 beats per minute (bpm), QTc interval less than or equal to (<=) 450 milliseconds (ms) for males, <=470 for females, QRS interval of less than (<) 120 ms, PR interval <210 ms, Morphology consistent with healthy cardiac conduction and function

Exclusion Criteria:

* Known allergies to seltorexant, zolpidem, and suvorexant
* Previous history of recurrent fainting, collapses, syncope, orthostatic hypotension, or vasovagal reactions
* Prescription medications except for stable medical problems such as hypertension, elevated cholesterol, and non-insulin-dependent diabetes mellitus with stable medications for at least 1 month prior to screening
* Participants who have ever been in treatment for substance use disorders (except smoking cessation) or are currently seeking treatment for substance use disorders. In addition, currently seeking or participating in a substance rehabilitation program should be excluded
* Preplanned surgery or procedures that would interfere with the conduct of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Peak Maximum Effect (Emax) for Drug Liking (At this Moment) Visual Analog Scale (VAS) | Up to 24 hour post-dose (up to Day 2)
  Emax for drug liking VAS will be reported. Drug liking VAS is a bipolar scale designed to assess a participant's liking for a given study intervention at the time the question is being asked (that is, at this moment). It is scored as an integer ranging from 0 (strong disliking) to 100 (strong liking).

SECONDARY OUTCOMES:
Overall Drug Liking VAS (Emax) | 12 hour and 24 hour post-dose
  Emax for overall drug liking VAS will be reported. Peak effect for overall drug liking based on bipolar VAS from 0 (strong disliking) to 100 (strong liking).
Take Drug Again VAS (Emax) | 12 hour and 24 hour post-dose
  Emax for take drug again VAS will be reported. Peak effect for take drug again based on bipolar VAS from 0 (definitely no) to 100 (definitely so).
Subjective Drug Value (Emax) | 12 hour and 24 hour post-dose
  Subjective drug value will be reported. The subjective drug value is a proxy measure of reinforcing efficacy that involves a series of independent, theoretical forced choices between drug administered and different monetary values.
High VAS (Emax) | Pre-dose up to 24 hours post-dose (up to Day 2)
  High VAS is one of the measures of positive effects that assesses the effect experienced by the participant on a 100 millimeter (mm) unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 = definitely so).
Time to Peak Effect (TEmax) for Drug Liking (At this Moment) VAS | Up to 24 hour post-dose (up to Day 2)
  TEmax is defined as time to peak effect for drug liking (at this moment). Drug liking VAS is a bipolar scale designed to assess a participant's liking for a given study intervention at the time the question is being asked (that is, at this moment). It is scored as an integer ranging from 0 (strong disliking) to 100 (strong liking).
Minimum Effect (Emin) for Drug Liking (At this Moment) VAS | Up to 24 hour post-dose (up to Day 2)
  Emin is defined as minimum effect for drug liking (at this moment). Drug liking VAS is a bipolar scale designed to assess a participant's liking for a given study intervention at the time the question is being asked (that is, at this moment). It is scored as an integer ranging from 0 (strong disliking) to 100 (strong liking).
Time to Minimum Effect (TEmin) for Drug Liking (At this Moment) VAS | Up to 24 hour post-dose (up to Day 2)
  TEmin is defined as time to minimum effect for drug liking (at this moment). Drug liking VAS is a bipolar scale designed to assess a participant's liking for a given study intervention at the time the question is being asked (that is, at this moment). It is scored as an integer ranging from 0 (strong disliking) to 100 (strong liking).
Time-averaged Area Under the Effects Curve (TA_AUE) for Drug Liking (At This Moment) VAS | Up to 24 hour post-dose (up to Day 2)
  TA_AUE is defined as time-averaged area under the effects curve for drug liking (at this moment). Drug liking VAS is a bipolar scale designed to assess a participant's liking for a given study intervention at the time the question is being asked (that is, at this moment). It is scored as an integer ranging from 0 (strong disliking) to 100 (strong liking).
TEmax of High VAS | Pre-dose up to 24 hours post-dose (up to Day 2)
  TEmax of high VAS will be reported. High VAS is one of the measures of positive effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 = definitely so).
TA_AUE of High VAS | Pre-dose up to 24 hours post-dose (up to Day 2)
  TA_AUE of high VAS will be reported. High VAS is one of the measures of positive effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 = definitely so).
Emax of Good Effect VAS | Up to 24 hour post-dose (up to Day 2)
  Emax of good effect VAS will be reported. Good drug effects VAS is one of the measures of positive effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 mm= definitely so).
TEmax of Good Effects VAS | Up to 24 hour post-dose (up to Day 2)
  TEmax of good effects VAS will be reported. Good drug effects VAS is one of the measures of positive effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 mm= definitely so).
TA_AUE of Good Effects VAS | Up to 24 hour post-dose (up to Day 2)
  TA_AUE of good effects VAS will be reported. Good drug effects VAS is one of the measures of positive effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 mm= definitely so).
Emax of Bad Effects VAS | Up to 24 hour post-dose (up to Day 2)
  Emax of bad effects VAS will be reported. Bad effects VAS measures the negative effects experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (0 mm = 'definitely not') to 'extremely' (100 mm = 'definitely so').
TA_AUE of Bad Effects VAS | Up to 24 hour post-dose (up to Day 2)
  TA_AUE for bad effects VAS will be reported. Bad effects VAS measures the negative effects experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (0 mm = 'definitely not') to 'extremely' (100 mm = 'definitely so').
TEmax of Bad Effects VAS | Up to 24 hour post-dose (up to Day 2)
  TEmax of bad effects VAS will be reported. Bad effects VAS measures the negative effects experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (0 mm = 'definitely not') to 'extremely' (100 mm = 'definitely so').
Emin of Drowsiness/Alertness VAS | Pre-dose up to 24 hours post-dose (up to Day 2)
  Emin of Drowsiness/Alertness VAS will be reported. Alertness/Drowsiness VAS measures the sedative effects. It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of 'neither drowsy nor alert' (score of 50 mm), on the left with 'very drowsy' (score of 0 mm) and on the right with 'very alert' (score of 100 mm).
TEmin of Drowsiness/Alertness VAS | Pre-dose up to 24 hours post-dose (up to Day 2)
  TEmin of Drowsiness/Alertness VAS will be reported. Alertness/Drowsiness VAS measures the sedative effects. It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of 'neither drowsy nor alert' (score of 50 mm), on the left with 'very drowsy' (score of 0 mm) and on the right with 'very alert' (score of 100 mm).
Time-averaged Area Over the Effect Time Curve (TA_AOE) of Drowsiness/Alertness VAS | Pre-dose up to 24 hours post-dose (up to Day 2)
  TA_AOE is defined as time-averaged area over the effect time curve. Alertness/Drowsiness VAS measures the sedative effects. It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of 'neither drowsy nor alert' (score of 50 mm), on the left with 'very drowsy' (score of 0 mm) and on the right with 'very alert' (score of 100 mm).
Emin of Relaxation/Agitation VAS | Pre-dose up to 24 hours post-dose (up to Day 2)
  Emin of relaxation/agitation VAS will be reported. Agitation/Relaxation VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm).
TEmin of Relaxation/Agitation VAS | Pre-dose up to 24 hours post-dose (up to Day 2)
  TEmin of relaxation/agitation VAS will be reported. Agitation/Relaxation VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm).
TA_AOE of Relaxation/Agitation VAS | Pre-dose up to 24 hours post-dose (up to Day 2)
  TA_AOE of relaxation/agitation VAS will be reported. Agitation/Relaxation VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm).
TEmax of Dizziness VAS | Pre-dose up to 24 hour post-dose (up to Day 2)
  TEmax of dizziness VAS will be reported. Dizziness VAS assesses the effect of dizziness by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm).
Emax of Dizziness VAS | Pre-dose up to 24 hour post-dose (up to Day 2)
  Emax of dizziness VAS will be reported. Dizziness VAS assesses the effect of dizziness by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm).
TA_AUE of Dizziness VAS | Pre-dose up to 24 hour post-dose (up to Day 2)
  TA_AUE of dizziness VAS will be reported. Dizziness VAS assesses the effect of dizziness by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm).
Emax of Any Effects VAS | Up to 24 hour post-dose (up to Day 2)
  Emax of any effects VAS will be reported. Any drug effects VAS measures other subjective effects experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (0 mm = 'definitely not') to 'extremely' (100 mm = 'definitely so').
TEmax of Any Effects VAS | Up to 24 hour post-dose (up to Day 2)
  TEmax of any effects VAS will be reported. Any drug effects VAS measures other subjective effects experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (0 mm = 'definitely not') to 'extremely' (100 mm = 'definitely so').
TA_AUE of Any Effects VAS | Up to 24 hour post-dose (up to Day 2)
  TA_AUE of any effects VAS will be reported. Any drug effects VAS measures other subjective effects experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (0 mm = 'definitely not') to 'extremely' (100 mm = 'definitely so').
Drug Similarity VAS | 24 hour post-dose
  Drug similarity VAS will be reported. The Drug Similarity unipolar VAS items provide an estimate of the drug class with which drug users identify the test drug. It is a unipolar scale ranging from 0 (not at all similar) to 100 points ( very similar).
Percentage of Participants with Adverse Events (AEs) | Up to Week 20
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Percentage of Participants with Serious Adverse Events (SAEs) | Up to Week 20
  An SAE is defined as any untoward medical occurrence that: results in death, is life-threatening, requires in patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, or is an important medical event.
Percentage of Participants with Abnormalities in Clinical Laboratory Parameters | Up to 24 hour post-dose (up to Day 2)
  Percentage of participants with abnormalities in clinical laboratory parameters (included hematology, clinical chemistry, and routine urinalysis) will be reported.
Percentage of Participants with Abnormalities in Vital Signs | Up to 24 hour post-dose (up to Day 2)
  Percentage of participants with abnormalities in vital signs (included temperature, pulse/heart rate, blood pressure [diastolic and systolic]) will be reported.
Emin of Modified Observer's Assessment of Alertness/Sedation (MOAA/S) of Composite and Sum Score | Up to 24 hour post-dose (up to Day 2)
  Emin of MOAA/S of composite and sum score will be reported. The MOAA/S is an observer-rated measure of alertness/sedation that is used widely in clinical research. The MOAA/S scores range from 5 (not sedated) to 0 (unarousable). The observer's assessment of alertness/sedation scale (OAA/S) was developed to measure the level of alertness in participants who are sedated. The OAA/S is a reliable validated measure and was shown to be sensitive to different levels of sedation and is composed of 4 assessment categories that include responsiveness, speech, facial expression, and eyes. The MOAA/S includes only the Responsiveness assessment category.
TA_AOE of MOAA/S of composite and sum score | Up to 24 hour post-dose (up to Day 2)
  TA_AOE of MOAA/S of composite and sum score will be reported. The MOAA/S is an observer-rated measure of alertness/sedation that is used widely in clinical research. The MOAA/S scores range from 5 (not sedated) to 0 (unarousable). The observer's assessment of alertness/sedation scale (OAA/S) was developed to measure the level of alertness in participants who are sedated. The OAA/S is a reliable validated measure and was shown to be sensitive to different levels of sedation and is composed of 4 assessment categories that include responsiveness, speech, facial expression, and eyes. The MOAA/S includes only the Responsiveness assessment category.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Altasciences Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency